CLINICAL TRIAL: NCT06486376
Title: The Impact of Teacher-led School Based Hygiene Campaign on Handwashing Practices and Prevention of Diarrhoea, Undernutrition and Pneumonia Among School Children in Nigeria.
Brief Title: The Impact of WASH on Handwashing Practices Among School Children in Nigeria.
Acronym: WASHEDUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Neo Child Initiative for Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-24-011
Record Dates: First submitted 2024-06-22; First posted 2024-07-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hand Hygiene
Keywords: WASH, schools, children
MeSH Terms: interventions — Water; Sanitation

STUDY DESIGN:
Intervention Model Description: School Cluster randomized trial study of 50 schools
Who Masked: Outcomes Assessor
Masking Description: The intervention is WASHED-UP (Water, Sanitation and Hygiene Education Against Diarrhoea, Undernutrition and Pneumonia), a 2-week health awareness campaign that will train children and teachers to deliver the program on hygiene promotion in schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active comparator (Active Comparator): Control Group: These will be schools where no intervention will be implemented, and routine practices are continued.
  Interventions: Behavioral: Water, Sanitation and Hygiene Education Against Diarrhoea, Undernutrition and Pneumonia
- Control (No Intervention): No intervention group

INTERVENTIONS:
Behavioral: Water, Sanitation and Hygiene Education Against Diarrhoea, Undernutrition and Pneumonia — Intervention components include teacher training, stepdown training of teachers to children and distribution of IEC materials.
  Other Names: WASHED-UP
  Arms: Active comparator

SUMMARY:
Children are considered as the most vulnerable group of individuals affected by lack of water, sanitation and hygiene facilities which predisposes them to a wide range of enteric diseases particularly diarrhoeal and parasitic infections. School-based WASH interventions typically aim to reduce the incidence of hygiene related diseases, improve school outcomes for pupils and influence hygiene practices of families and the wider community. This study intends to investigate the impact and effectiveness of the teacher-led school- based hygiene intervention on handwashing practices and prevention of diarrhoea, undernutrition, and pneumonia among school children in primary schools in Lagos, Nigeria.

DETAILED DESCRIPTION:
This research project will be conducted as a school cluster-randomized study with 50 randomly selected low-cost private primary schools in the Lagos region. The expected number of schools included is 25 intervention and 25 control schools (schools that have not received the intervention but that are similar enough to the intervention schools to facilitate comparison). Quantitative data will be collected on the implementation and impact of the intervention, and qualitative data will be collected to explore teacher perceptions of best WASH practices. The intervention WASHED-UP (Water, Sanitation and Hygiene Education Against Diarrhoea, Undernutrition and Pneumonia) will be implemented as a 2-week health awareness campaign that will train children and teachers to deliver the program on hygiene promotion in schools. Intervention components include the presentation of interactive stories, games and songs, nutrition education, participatory food demonstration classes using food models, the use of animated characters representing occasions for handwashing with soap, practical and visual demonstrations to communicate the presence of germs and handwashing with soap removes them in comparison to only water, the use of daily diaries by students to record their handwashing behaviour and making a public commitment to handwashing with soap as a club. Digital surveys and implementation checklists will be used to collect the impact (survey) and implementation data, respectively and audio recordings of focus groups will be used to collect data related to stakeholder perceptions of the WASHED-UP program. For school absence, data are planned to be obtained from paper-based school records, including registers and sick-bay records. Approximately 3500 children will be recruited for data collection which will involve administering questions on socio-demographics, illness, reasons for school absence, disease history, sanitation behaviour at home and school and attendance at WASH clubs. At the end of the study all control schools will receive the intervention subsequently.

Data will be collected in three phases:

* Phase 1: February to March 2024 and will consist of a baseline survey.
* Phase 2: May to June 2024 and will consist of an implementation phase in the form of the intervention in the randomly selected 25 primary schools in Lagos.
* Phase 3: September to November 2024 and will consist of three months of follow-up post-implementation and comparison to control schools. Data will be collated using the Kobo Toolbox survey tool and analyzed with Statistical Package for Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Schools are located in Lagos state
* Schools must have functional WASH facilities:
* Schools must have access to a water source
* Schools have school registers

Exclusion Criteria:

* School authorities refuse to participate
* Schools which have received WASH intervention

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3500 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Sanitation and hygiene-related knowledge, attitudes, and practices of handwashing | 3 months
  The incidence of diarrhoeal diseases and pneumonia among school children in primary schools in Lagos.

SECONDARY OUTCOMES:
School absenteeism | 3 months
  The difference in school absence and the occurrence of self-reported diarrhoea, and pneumonia symptoms between children who attended schools that participated in the WASHED-UP campaign versus children who attended schools that did not receive WASHED-UP?

CONTACTS AND LOCATIONS:
Locations (1):
- Kiddies Primary School, Somolu, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Essential Study protocol and data collection tools will be shared with other researchers
Supporting Information: Study Protocol, ICF
Time Frame: June to December 2024